CLINICAL TRIAL: NCT04173195
Title: Comfort Talk (CT) to Improve Emotional Support and Physical Comfort During Outpatient Chemotherapy: a Pilot Study
Brief Title: Comfort Talk (CT) During Outpatient Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Caroline Arbour, Regular researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-1751
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Chemotherapy Effect
Keywords: Comfort talk; Outpatient clinic; Emotional support; Pain; Nursing care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This pilot trials will be conducted simultaneously in two outpatient oncology clinics located in the Montreal area: 1) Hôpital du Sacré-Coeur de Montréal, and 2) Hôpital de Saint-Eustache. These sites have been selected has they share the same hemato-oncologists, ensuring some consistency in treatment protocols. Site 1 will serve as the experimental site (combining CT with current care) and site 2 will serve as the control site (current care only).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will be blinded to treatment allocation. Complete blinding of care providers will not possible as the nurses in charge of chemotherapy admnistration will also be responsible to provide the CT intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The CT intervention will be administered by the nurse in charge of the chemotherapy 5 min after the initiation. the CT content will be partially script.
  Interventions: Other: Comfort Talk
- No intervention arm (No Intervention): Patients assigned to this arm will received current care.

INTERVENTIONS:
Other: Comfort Talk — A short and brief conversation based on the principles of clinical hypnosis.
  Arms: Intervention arm

SUMMARY:
Emotional support and physical comfort are two important components of the patient experience at the oncology outpatient clinic. However, current practices do not seem optimal for meeting the psychosocial needs expressed by patients during chemotherapy treatments.

Comfort talk (CT) is a simple, inexpensive intervention that could maximize the feeling of safety and comfort during chemotherapy. Identifying interventions that are interdisciplinary and that can enhance the outpatient patient experience will facilitate access to quality oncology care.

DETAILED DESCRIPTION:
The number of cancer cases requiring chemotherapy is on the rise in North America. About 84% of chemotherapy treatments are administered by nurses in a outpatient clinic context. Although outpatient oncology care are generally associated with a significant improvement in the quality of life in cancer patients, one-third of patients believe that health professionals (including nurses) are not doing everything in their power to comfort or relieve discomfort during chemotherapy treatments. Among the known elements for enhancing the well-being of oncology outpatients, comfort talk (CT) has been found to be very effective. Indeed, CT is a simple and direct form of conversation that is inspired by the principles of clinical hypnosis. While the soothing mechanisms of CT are poorly understood, involvement of cortical regions involved in the modulation of emotions and pain is suggested in several neuroimaging studies.This pilot trial serves as a proof of concept and aims to explore whether CT can be used by nurses to optimize the perception of emotional support and physical comfort during outpatient chemotherapy treatments. To do this, patients enrolled in a chemotherapy treatment cycle will be recruited during a visit to the oncology outpatient clinic. Half of the patients will be assigned to enhanced routine care with an CT intervention and the other half will receive routine care without CT. If there is an overlap between CT mechanisms and those involved in the endogenous control of emotions and pain, a significant interaction of these elements on the well-being of patients during chemotherapy treatments is expected. The results of this pilot trials will be used to justify and prepare for a larger study to evaluate the effects of CT on cancer symptom management and treatment at the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age and older) with cancer (regardless of stage) who have initiated a outpatient chemotherapy treatment cycle for at least 1 week and who are expected to receive at least two additional treatments related to this cycle will be considered for eligibility.

Exclusion Criteria:

* BMI ≥30 or pregnancy;
* With a history of pre-existing chronic pain;
* History of psychosis or serious mental illness;
* Receiving anti-cancer treatments for more than 2 years;
* Any other conditions that make the patient's participation potentially detrimental to his well-being as recommended by the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in emotional support | Immediately before/after CT
  Perceived support scale, 9 items rated on 0-100mm VAS, with 0 meaning that the support is completely absent and 100 that it is at its optimal level.
Changes in physical comfort | Immediately before/after CT
  Edmonton Symptom Assessment Scale, 9 items rated on 0-100mm VAS, with 0 meaning that the symptom is absent and 100 that it is the worst possible severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbour C, Tremblay M, Ogez D, Martineau-Lessard C, Lavigne G, Rainville P. Feasibility and acceptability of hypnosis-derived communication administered by trained nurses to improve patient well-being during outpatient chemotherapy: a pilot-controlled trial. Support Care Cancer. 2022 Jan;30(1):765-773. doi: 10.1007/s00520-021-06481-6. Epub 2021 Aug 10. PMID 34374847